CLINICAL TRIAL: NCT05835011
Title: A Phase 2 Study of Oral Decitabine/Cedazuridine in Combination With Magrolimab for Previously Untreated Subjects With Intermediate- to Very High-Risk Myelodysplastic Syndromes (MDS)
Brief Title: A Study of Oral Decitabine/Cedazuridine in Combination With Magrolimab in Participants With Intermediate- to Very High-Risk Myelodysplastic Syndromes (MDS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Termination due to discontinuation of magrolimab development in MDS.
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASTX727-10; 2022-501548-14-00 (Other: EU CTIS Number)
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Results first posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — decitabine and cedazuridine drug combination; magrolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oral Decitabine/Cedazuridine + Magrolimab (Experimental): Participants will receive 35 milligrams (mg) decitabine/100 mg cedazuridine as a fixed dose combination (FDC) tablet, orally, once daily (QD) on Days 1-5 of each 28-day cycle in combination with magrolimab, intravenous (IV) infusion of 1 milligrams per kilogram (mg/kg) on Days 1 and 4, 15 mg/kg on Day 8, 30 mg/kg on Days 11, 15, 22, 29, 36, 43, and 50, followed by a maintenance dose of 30 mg/kg on Day 57 and every 14 days thereafter until toxicity, progressive disease, withdrawal, death or end of study (approximately 44 months).
  Interventions: Drug: Decitabine/Cedazuridine; Drug: Magrolimab

INTERVENTIONS:
Drug: Decitabine/Cedazuridine — Oral FDC tablets administration
  Other Names: ASTX727; INQOVI
Drug: Magrolimab — IV administration
  Other Names: Hu5F9-G4

SUMMARY:
The primary purpose of the study is to evaluate the preliminary safety and efficacy of oral decitabine/cedazuridine in combination with magrolimab.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmation of previously untreated MDS (i.e., no hypomethylating agent [HMA], chemotherapy, or allogenic stem cell transplant [SCT] per World Health Organization 2016 classification with <20% bone marrow (BM) blasts per marrow biopsy/aspirate at screening.
2. Projected life expectancy of at least 3 months.
3. Overall Revised International Prognostic Scoring System for myelodysplastic syndromes (IPSS-R) score ≥3.5 MDS (immediate risk or higher).
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of ≤2.
5. Hematopoietic stem cell transplant (HSCT) eligible without any pre-arranged HSCT on Cycle 1 Day 1, or HSCT ineligible.
6. Blood type and screen (any of the 4 blood groups A, B, AB, and O [ABO]/rhesus factor [Rh]) along with extended red blood cell phenotyping or genotyping completed prior to study drug treatment.
7. Hemoglobin ≥9 grams per deciliter (g/dL) on the first day of drug administration, transfusions allowed.
8. Willing to undergo blood transfusions as per parameters of protocol and clinically necessary.
9. White blood cell count ≤20×103/microliters (μL) prior to first dose and throughout study. Hydroxyurea could have been used to achieve this goal prior to and during the first 56 days of magrolimab administration.

Exclusion Criteria:

- Medical Conditions:

1. Known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive), or hepatitis C (e.g., hepatitis C virus ribonucleic acid [HCV RNA] is detected), or chronic hepatitis B or C infection or human immunodeficiency virus (HIV) infection in medical history, with the following exceptions:

   1. Those with a history of hepatitis with a negative polymerase chain reaction (either qualitative or quantitative) OR have documentation of stable disease with aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase and alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase <2.0×upper limit of normal (ULN) may be eligible for this study.
   2. Participants with history of HIV who have an undetectable viral load for the prior 3 months, and who agree to maintain antiviral therapy, may be eligible for the study.
2. Significant medical diseases or conditions, as assessed by the investigators and sponsor, that would substantially increase the risk benefit ratio of participating in the study. This includes, but is not limited to, acute myocardial infarction within the last 6 months, unstable angina, uncontrolled diabetes mellitus, significant active infections, and congestive heart failure New York Heart Association Class III-IV.
3. Known inherited or acquired bleeding disorders that require medication or medical intervention.
4. Second malignancy, except treated basal cell or localized squamous skin carcinomas, localized prostate cancer, or other malignancies for which participants are not on active anticancer therapies and have had no evidence of active malignancy for at least ≥1 year.

   -Prior/Concomitant Therapy:
5. Immediate eligibility for an allogeneic SCT, as determined by the investigator, with an available donor.
6. Prior therapy for MDS with chemotherapy, allogenic SCT, or ≥1 full cycle of treatment with any HMA.
7. History of therapy-related MDS, MDS evolving from a pre-existing myeloproliferative neoplasm (MPN), MDS/MPN including chronic myelomonocytic leukemia (CMML), atypical chronic myeloid leukemia, juvenile myelomonocytic leukemia, and unclassifiable MDS/MPN.
8. Prior anti-cluster of differentiation 47 (CD47) treatment.
9. Previous SCT within 6 months before first dose administration, active graft-versus-host disease, or requiring transplant-related immunosuppression.

   -Other Exclusions:
10. Known or suspected hypersensitivity to decitabine, cedazuridine, magrolimab, or any of their excipients.
11. Known significant mental illness or other condition such as active alcohol or other substance abuse or addiction that, in the opinion of the investigator, predisposes the participant to high-risk of noncompliance with the protocol.
12. Clinical suspicion of active central nervous system (CNS) involvement by MDS.
13. History of psychiatric illness or substance abuse likely to interfere with the ability to comply with protocol requirements or give informed consent.
14. Pregnant or actively breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-06-27 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Yale University, New Haven, Connecticut
  - BRCR Medical Center, Plantation, Florida
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2 participants were enrolled at 2 sites in the United States.
Pre-assignment Details: Out of 2 enrolled participants, only 1 received treatment.
Groups:
- Oral Decitabine/Cedazuridine + Magrolimab: Participants were to receive 35 milligrams (mg) decitabine/100 mg cedazuridine as a fixed dose combination (FDC) tablet, orally, once daily (QD) on Days 1-5 of each 28-day cycle in combination with magrolimab, intravenous (IV) infusion of 1 milligrams per kilogram (mg/kg) on Days 1 and 4, 15 mg/kg on Day 8, 30 mg/kg on Days 11, 15, 22, 29, 36, 43, and 50, followed by a maintenance dose of 30 mg/kg on Day 57 and every 14 days thereafter until toxicity, progressive disease, withdrawal, death or end of study.
Period: Overall Study
Arm/Group | Oral Decitabine/Cedazuridine + Magrolimab
Started | 2
Completed | 0
Not Completed | 2
Not completed — Study Terminated by the Sponsor | 1
Not completed — Enrolled but did not receive study treatment | 1

BASELINE CHARACTERISTICS:
Population: The study was terminated by the Sponsor. Based on the low enrollment number (n=2), no data, except region of enrollment, is reported here to protect and maintain participant privacy/confidentiality.
Groups:
- Oral Decitabine/Cedazuridine + Magrolimab: Participants were to receive 35 mg decitabine/100 mg cedazuridine as a FDC tablet, orally, QD on Days 1-5 of each 28-day cycle in combination with magrolimab, IV infusion of 1 mg/kg on Days 1 and 4, 15 mg/kg on Day 8, 30 mg/kg on Days 11, 15, 22, 29, 36, 43, and 50, followed by a maintenance dose of 30 mg/kg on Day 57 and every 14 days thereafter until toxicity, progressive disease, withdrawal, death or end of study.
Arm/Group | Oral Decitabine/Cedazuridine + Magrolimab
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The study was terminated by the Sponsor. Based on the low enrollment number (n=2), no data is reported here to protect and maintain participant privacy/confidentiality.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The study was terminated by the Sponsor. Based on the low enrollment number (n=2), no data is reported here to protect and maintain participant privacy/confidentiality.
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The study was terminated by the Sponsor. Based on the low enrollment number (n=2), no data is reported here to protect and maintain participant privacy/confidentiality.
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The study was terminated by the Sponsor. Based on the low enrollment number (n=1), no data is reported here to protect and maintain participant privacy/confidentiality.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) Graded According to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0
Description: An AE is any untoward medical occurrence in a subject or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention.
Time Frame: From signing of informed consent to 30 days after last dose of study drug (Up to 8 weeks)
Population: The safety population included the participant who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Decitabine/Cedazuridine + Magrolimab
Number analyzed (Participants) | 1
Participants | 1

2. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: DLTs are defined as any of the following toxicities at least possibly related to the treatment regimen: drug-related Grade ≥3 non-hematologic event; grade 4 neutropenia and thrombocytopenia that was not present prior to dosing, that last 28 days or longer and is not related to underlying disease; or any drug-related toxicity that result in treatment delay of >2 weeks after Cycle 1 (28 days) is complete.
Time Frame: From signing of informed consent to 30 days after last dose of study drug (Up to 8 weeks)
Population: The safety population included participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Decitabine/Cedazuridine + Magrolimab
Number analyzed (Participants) | 1
Participants | 0

3. Primary Outcome: Complete Response (CR) Rate
Description: CR defined as per International Working Group (IWG) criteria 2006: Bone marrow (BM) ≤5% myeloblasts with normal maturation of all cell lines; Persistent dysplasia; Peripheral blood; Hemoglobin (Hgb) ≥11 g/dL; Platelets ≥100×109/L; Neutrophils ≥1.0×109/Lb; Blasts 0%. Per the response criteria the response must last ≥4 weeks.
Time Frame: Up to 44 months
Population: As pre-specified in the protocol, analysis of the CR rate was to be conducted 8 months after the enrollment of approximately 100 participants in the study. As only 1 participant received study drug, hence no data was collected for this outcome measure.
Arm/Group | Oral Decitabine/Cedazuridine + Magrolimab
Number analyzed (Participants) | 0

4. Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) of Oral Decitabine/Cedazuridine and Magrolimab
Time Frame: Decitabine/Cedazuridine: Multiple timepoints pre-dose and post dose up to Day 5 of Cycle 1 and Day 4 of Cycle 2 (Cycle=28 days); Magrolimab: Multiple timepoints pre-dose and post dose up to end of treatment (up to 44 months)
Population: Data for this outcome measure was not collected and analyzed as planned as the study was terminated due to discontinuation of magrolimab development in MDS.
Arm/Group | Oral Decitabine/Cedazuridine + Magrolimab
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as percentage of participants with CR, partial response (PR), marrow complete response (mCR), and hematologic improvement (HI). CR: Bone marrow (BM) ≤5% myeloblasts with normal maturation of all cell lines; Persistent dysplasia; Peripheral blood; Hemoglobin (Hgb) ≥11 g/dL; Platelets ≥100×109/L; Neutrophils ≥1.0×109/Lb; Blasts 0%. PR: all CR criteria if abnormal before treatment except: BM blasts decreased by ≥50% over pretreatment but still >5%; cellularity and morphology not relevant. mCR: BM ≤5% myeloblasts and decrease by ≥50% over pretreatment; peripheral blood- if HI responses, they are noted in addition to marrow CR. HI include HI with Erythroid (HI-E), HI with Neutrophil (HI-N), or HI with Platelet (HI-P). Per the response criteria the response must last ≥4 weeks for CR, PR and mCR. For HI, the response must last ≥8 weeks.
Time Frame: Up to 44 months
Population: As only 1 participant received study drug, data for this outcome measure was not collected and analyzed as planned as the study was terminated due to discontinuation of magrolimab development in MDS.
Arm/Group | Oral Decitabine/Cedazuridine + Magrolimab
Number analyzed (Participants) | 0

6. Secondary Outcome: Rate of Hematologic Improvement (HI)
Description: HI include HI-E, HI-N, or HI-P based on the 2006 International Working Group Criteria (IWG 2006). HI-E: Hemoglobin (Hgb) increase ≥1.5g/dL, Relevant reduction of red blood cell (RBC) units transfusions by absolute ≥4 RBC transfusions/8 week compared with pretreatment transfusion number previous 8 week. Only RBC transfusions given for Hgb ≤9.0 g/dL. HI-P: Absolute increase ≥30x10^9/L starting >20x10^9/L platelets (PLTs); Increase from <20x10^9/L to >20x10^9/L and by≥100%. HI-N: ≥100% increase, absolute increase>0.5x10^9/L. Per the response criteria the response must last ≥8 weeks.
Time Frame: Up to 44 months
Population: as for outcome 5
Arm/Group | Oral Decitabine/Cedazuridine + Magrolimab
Number analyzed (Participants) | 0

7. Secondary Outcome: Duration of Progression Free Survival (PFS)
Description: PFS is defined as time from the date of randomization to the date of disease progression. Disease progression is: For participants with less than 5% blasts: ≥50 increase in blasts to >5% blasts; 5%-10% blasts: ≥50% increase in blasts to >10% blasts; 10%-20% blasts: ≥50% increase in blasts to >20% blasts; 20%-30% blasts: ≥50% increase in blasts to >30% blasts and any of the following: at least 50% decrement from maximum remission/response in granulocytes or platelets; Reduction in Hgb by ≥2 g/dL; transfusion dependence. Per the response criteria the response must last ≥4 weeks.
Time Frame: Up to 44 months
Population: as for outcome 5
Arm/Group | Oral Decitabine/Cedazuridine + Magrolimab
Number analyzed (Participants) | 0

8. Secondary Outcome: Leukemia-free Survival (LFS)
Description: LFS is defined as the number of days from date of randomization to date when bone marrow or peripheral blood blasts reach ≥20%, or death.
Time Frame: Up to 44 months
Population: as for outcome 5
Arm/Group | Oral Decitabine/Cedazuridine + Magrolimab
Number analyzed (Participants) | 0

9. Secondary Outcome: Percentage of Participants With Minimal Residual Disease (MRD)-Negative Status
Time Frame: Day 1 of each 28-day Cycle starting from Cycle 3 up to end of study (up to 44 months)
Population: Before Cycle 3 was initiated for 1 participant who received study drug, the study was prematurely terminated due to discontinuation of magrolimab development in MDS. Hence, no data was collected for this outcome
Arm/Group | Oral Decitabine/Cedazuridine + Magrolimab
Number analyzed (Participants) | 0

10. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from the date that measurement criteria are first met for CR or PR until the first subsequent date that progressive disease or death is documented.
Time Frame: Up to 44 months
Population: as for outcome 5
Arm/Group | Oral Decitabine/Cedazuridine + Magrolimab
Number analyzed (Participants) | 0

11. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as time from the date of randomization to the date of death from any cause.
Time Frame: Up to 44 months
Population: as for outcome 5
Arm/Group | Oral Decitabine/Cedazuridine + Magrolimab
Number analyzed (Participants) | 0

12. Secondary Outcome: Number of Participants With International Prognostic Scoring System for Myelodysplastic Syndromes (IPSS-M) Score
Description: The IPSS-M is an algorithm that uses clinical features of participants with MDS and assigns a prognostic score (0=good and increasing in risk by half-grades with the top score outlined below) for three prognostic variables: Marrow blasts (score 0-2.0); Karyotype (score 0-1.0); Cytopenias: neutrophil, platelets, and Hg counts (score 0-0.5). The three individual scores are summed resulting in a full range of 0- 3.5 and placed into risk categories: 0 = low risk; 0.5-1.0 = intermediate-1 risk; 1.5-2.0 = intermediate-2 risk; and >=2.5 = high risk. Higher scores indicate worst outcome.
Time Frame: Up to Day 42
Population: as for outcome 5
Arm/Group | Oral Decitabine/Cedazuridine + Magrolimab
Number analyzed (Participants) | 0

13. Secondary Outcome: Number of Participants With p53 Mutation
Time Frame: Up to Day 42
Population: as for outcome 5
Arm/Group | Oral Decitabine/Cedazuridine + Magrolimab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From signing of informed consent to 30 days after last dose of study drug (Up to 8 weeks)
Description: The safety population included the participant who received at least one dose of study treatment.
Arm/Group | Oral Decitabine/Cedazuridine + Magrolimab
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Decitabine/Cedazuridine + Magrolimab (N=1)
Platelet count decreased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Intermittent dizziness (Nervous system disorders) | 1 (1)
Intermittent anaemia (Blood and lymphatic system disorders) | 1 (1)
Intermittent platelet count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated prematurely due to discontinuation of magrolimab development in MDS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-19): https://cdn.clinicaltrials.gov/large-docs/11/NCT05835011/Prot_SAP_000.pdf